CLINICAL TRIAL: NCT06756477
Title: The Effect of Mindfulness-Based Healthy Living Behaviors Training on Premenstrual Syndrome Symptoms and Quality of Life
Brief Title: The Effect of Mindfulness Training on Premenstrual Syndrome Symptoms and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nisan Akçay (Other)
Responsible Party: Sponsor-Investigator, Nisan Akçay, specialized midwife, Gulhane School of Medicine
Organization: Gulhane School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: nisanakçay00001
Record Dates: First submitted 2024-12-21; First posted 2025-01-03 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Mindfulness; Premenstrual Syndrome-PMS; Quality of Life
Keywords: Mindfulness-Based Education; Healthy Living Behaviours; Premenstrual Syndrome Symptoms; Quality of Life; Midwifery
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): Mindfulness group
  Interventions: Behavioral: mindfulness group; Other: control group
- Control (No Intervention): standard training group

INTERVENTIONS:
Behavioral: mindfulness group — Online training will be implemented 2 times a week for 8 sessions. A 30-45 minute reminder training will be given 1 month after the training. Mindfulness-Based Healthy Living Behaviors Education (MTSYDE) booklet will be sent online to guide students' home practices. Taking into account the possibility of forgetting and demotivation in students, audio recordings will be used, reminder messages will be sent and counseling will be given regarding the program. A post-test will be administered 1 month after the reminder training.
  Arms: Mindfulness
Other: control group — Menstruation-specific Healthy Living Behaviors training of 30-45 minutes in 8 sessions 2 times a week will be provided online. A standard training booklet will be sent 1 month after the training as a reminder. Standard reminder messages will be sent considering the possibility of forgetting and demotivation in students. A post-test will be administered 1 month after the reminder training.
  Arms: Mindfulness

SUMMARY:
Premenstrual syndrome (PMS) is an important health problem that negatively affects women's quality of life by reducing their daily activities, sleep quality, cognitive functioning, interpersonal relationships, academic performance, work and school attendance. Studies show that PMS is associated with unhealthy life behaviors and that PMS can be reduced through the development of healthy life behaviors. Midwives can benefit from mindfulness-based programs while providing quality health care services to develop a healthy lifestyle in the prevention and treatment of PMS in women. In the literature, there is no study examining the effectiveness of mindfulness-based healthy life behaviors training on PMS. To the best of our knowledge, our study is the first study to examine the effect of a mindfulness-based healthy life behaviors training program on premenstrual syndrome symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Regular menstruation Those who score at least 132 or higher on the PMS scale Agreeing to participate in the study With internet access

Exclusion Criteria:

Having a psychiatric diagnosis or gynecological disease Kontraseptif medication use Having a health problem Receiving treatment for PMS

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Having moderate symptoms of premenstrual syndrome
Enrollment: 114 (Actual)
Dates: Start 2025-05-03 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-08-03 (Actual)

PRIMARY OUTCOMES:
Premenstrual Syndrome Scale (PMSS) | Before the start of training and 2 months after the first training
  The total score ranges between 44-220. The higher the score, the higher the intensity of premenstrual syndrome symptoms.
Premenstrual syndrome-specific quality of life scale | Before the training and 2 months after the first training is completed
  The total score ranges from 22 to 110, with higher scores indicating better life behaviors.
Quality of Life Visual Analog Scale (VAS) | Before the training and 2 months after the first training is completed
  Total scale scores range from 0-10. The higher the scale scores, the better the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Çankaya Ilçe Sağlık Müdürlüğü, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dawson AF, Brown WW, Anderson J, Datta B, Donald JN, Hong K, Allan S, Mole TB, Jones PB, Galante J. Mindfulness-Based Interventions for University Students: A Systematic Review and Meta-Analysis of Randomised Controlled Trials. Appl Psychol Health Well Being. 2020 Jul;12(2):384-410. doi: 10.1111/aphw.12188. Epub 2019 Nov 19. PMID 31743957
- [Result] Yildirim Sisman N, Karaca A, Cangur S. Factors affecti̇ng health-promoting behavi̇ors i̇n nursi̇ng students: A structural equation modeling approach. Nurse Educ Pract. 2020 Oct;48:102880. doi: 10.1016/j.nepr.2020.102880. Epub 2020 Sep 1. PMID 32911210
- [Result] Kaisti I, Kulmala P, Hintsanen M, Hurtig T, Repo S, Paunio T, Miettunen J, Halt AH, Jaaskelainen E. The effects of mindfulness-based interventions in medical students: a systematic review. Adv Health Sci Educ Theory Pract. 2024 Mar;29(1):245-271. doi: 10.1007/s10459-023-10231-0. Epub 2023 May 25. PMID 37227541
- [Result] Jose A, Nayak S, Rajesh A, Kamath N, Nalini M. Impact of relaxation therapy on premenstrual symptoms: A systematic review. J Educ Health Promot. 2022 Dec 28;11(1):401. doi: 10.4103/jehp.jehp_586_22. eCollection 2022. PMID 36824400
- [Result] Yan H, Wu Y, Li H. Effect of mindfulness-based interventions on mental health of perinatal women with or without current mental health issues: A systematic review and meta-analysis of randomized controlled trials. J Affect Disord. 2022 May 15;305:102-114. doi: 10.1016/j.jad.2022.03.002. Epub 2022 Mar 4. PMID 35257692
- [Result] Wells RE, O'Connell N, Pierce CR, Estave P, Penzien DB, Loder E, Zeidan F, Houle TT. Effectiveness of Mindfulness Meditation vs Headache Education for Adults With Migraine: A Randomized Clinical Trial. JAMA Intern Med. 2021 Mar 1;181(3):317-328. doi: 10.1001/jamainternmed.2020.7090. PMID 33315046
- [Result] Valikhani A, Kashani VO, Rahmanian M, Sattarian R, Rahmati Kankat L, Mills PJ. Examining the mediating role of perceived stress in the relationship between mindfulness and quality of life and mental health: testing the mindfulness stress buffering model. Anxiety Stress Coping. 2020 May;33(3):311-325. doi: 10.1080/10615806.2020.1723006. Epub 2020 Feb 6. PMID 32026721
- [Result] Ibici Akca E, Gokbulut N, Cengizhan SO. The Effects of MBSR Programme on Prenatal Comfort and Fetal Health Anxiety in Pregnant Women. J Reprod Infant Psychol. 2024 Jun;42(3):449-463. doi: 10.1080/02646838.2023.2227219. Epub 2023 Jun 21. PMID 37342975
- [Result] Kundarti FI, Titisari I, Rahayu DE, Kiswati, Jamhariyah. Mindfulness improves the mental health of infertile women: A systematic review. J Public Health Res. 2023 Sep 12;12(3):22799036231196693. doi: 10.1177/22799036231196693. eCollection 2023 Jul. PMID 37711728
- [Result] Ni Y, Ma L, Li J. Effects of Mindfulness-Based Stress Reduction and Mindfulness-Based Cognitive Therapy in People With Diabetes: A Systematic Review and Meta-Analysis. J Nurs Scholarsh. 2020 Jul;52(4):379-388. doi: 10.1111/jnu.12560. Epub 2020 May 14. PMID 32406186
- [Result] Chen Q, Liu H, Du S. Effect of mindfulness-based interventions on people with prehypertension or hypertension: a systematic review and meta-analysis of randomized controlled trials. BMC Cardiovasc Disord. 2024 Feb 14;24(1):104. doi: 10.1186/s12872-024-03746-w. PMID 38350849
- [Result] Park S, Sato Y, Takita Y, Tamura N, Ninomiya A, Kosugi T, Sado M, Nakagawa A, Takahashi M, Hayashida T, Fujisawa D. Mindfulness-Based Cognitive Therapy for Psychological Distress, Fear of Cancer Recurrence, Fatigue, Spiritual Well-Being, and Quality of Life in Patients With Breast Cancer-A Randomized Controlled Trial. J Pain Symptom Manage. 2020 Aug;60(2):381-389. doi: 10.1016/j.jpainsymman.2020.02.017. Epub 2020 Feb 24. PMID 32105790
- [Result] Gordon JL, Halleran M, Beshai S, Eisenlohr-Moul TA, Frederick J, Campbell TS. Endocrine and psychosocial moderators of mindfulness-based stress reduction for the prevention of perimenopausal depressive symptoms: A randomized controlled trial. Psychoneuroendocrinology. 2021 Aug;130:105277. doi: 10.1016/j.psyneuen.2021.105277. Epub 2021 May 19. PMID 34058560
- [Result] Yazdani Aliabadi M, Javadnoori M, Saki Malehi A, Aslani K. A study of mindfulness-based stress-reduction training effects on menopause-specific quality of life in postmenopausal women: A randomized controlled trial. Complement Ther Clin Pract. 2021 Aug;44:101398. doi: 10.1016/j.ctcp.2021.101398. Epub 2021 Apr 24. PMID 33915368
- [Result] Mazaheri Asadi D, Zahedi Tajrishi K, Gharaei B. Mindfulness Training Intervention With the Persian Version of the Mindfulness Training Mobile App for Premenstrual Syndrome: A Randomized Controlled Trial. Front Psychiatry. 2022 Jun 17;13:922360. doi: 10.3389/fpsyt.2022.922360. eCollection 2022. PMID 35782413
- [Result] Solt Kirca A, Kizilkaya T. Effects of music medicine on premenstrual symptoms levels and quality of life: A randomized controlled trial. Complement Ther Clin Pract. 2022 Feb;46:101542. doi: 10.1016/j.ctcp.2022.101542. Epub 2022 Feb 5. PMID 35149373
- [Result] Ayaz-Alkaya S, Yaman-Sozbir S, Terzi H. The effect of Health Belief Model-based health education programme on coping with premenstrual syndrome: a randomised controlled trial. Int J Nurs Pract. 2020 Apr;26(2):e12816. doi: 10.1111/ijn.12816. Epub 2020 Jan 27. PMID 31985138
- [Result] Kwon YJ, Sung DI, Lee JW. Association among Premenstrual Syndrome, Dietary Patterns, and Adherence to Mediterranean Diet. Nutrients. 2022 Jun 14;14(12):2460. doi: 10.3390/nu14122460. PMID 35745189
- [Result] Jaber RM, Alghzawi AO, Salameh HH. Premenstrual syndrome: consultation sources and the impact on women's quality of life. Afr Health Sci. 2022 Mar;22(1):80-87. doi: 10.4314/ahs.v22i1.10. PMID 36032464
- [Result] Vieira AKS, Nagumo MT, Kuba G, Kurebayashi LFS, Turrini RNT. Effect of Foot Reflexology Protocol on Premenstrual Syndrome Symptoms in Nursing Students: a Pre-Post Pilot Study. Int J Ther Massage Bodywork. 2021 Dec 1;14(4):1-11. doi: 10.3822/ijtmb.v14i4.631. eCollection 2021 Dec. PMID 34900066
- [Result] Al-Shahrani AM, Miskeen E, Shroff F, Elnour S, Algahtani R, Youssry I, Ahmed S. Premenstrual Syndrome and Its Impact on the Quality of Life of Female Medical Students at Bisha University, Saudi Arabia. J Multidiscip Healthc. 2021 Aug 27;14:2373-2379. doi: 10.2147/JMDH.S327893. eCollection 2021. PMID 34475764
- [Result] Mushtaq A, Arif S, Sabih F. Premenstrual symptoms as predictor of quality of life in reproductive-aged women of Rawalakot, Azad Kashmir: A cross sectional study. J Pak Med Assoc. 2020 Dec;70(12(B)):2394-2397. doi: 10.47391/JPMA.417. PMID 33475550